CLINICAL TRIAL: NCT07221617
Title: Oral Methadone In Cardiac Surgery
Acronym: OMICS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Krishnan Ramanujan, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 25-007292
Record Dates: First submitted 2025-10-25; First posted 2025-10-28 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Pain, Postoperative; Anesthesia; Cardiac Surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Methadone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intravenous methadone intraoperatively (Active Comparator): Subjects in the IV methadone arm will receive methadone intravenously during cardiac surgery
  Interventions: Drug: Methadone, intravenously
- Oral methadone, immediately prior to transport (Experimental): Subjects in the oral methadone arm will receive methadone orally prior to cardiac surgery
  Interventions: Drug: Methadone, oral

INTERVENTIONS:
Drug: Methadone, oral — Patients will receive 0.4mg/kg PO methadone immediately prior to transport to the operating room
  Arms: Oral methadone, immediately prior to transport
Drug: Methadone, intravenously — Patients will receive 0.3mg/kg methadone intravenously after induction of general anesthesia
  Arms: Intravenous methadone intraoperatively

SUMMARY:
The purpose of this study is to compare the effects of administration of oral methadone preoperatively and intravenous methadone upon induction of general anesthesia on postoperative pain for patients undergoing elective cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

• Undergoing elective cardiac surgery

Exclusion Criteria:

* Chronic pain requiring opioid medications as an outpatient
* Opioid use disorder on medication assistance treatment
* Prolonged QTc >500ms
* Chronic kidney disease with eGFR < 30mL/min
* Documented cirrhosis
* Intolerance to methadone
* Admitted inpatient in an intensive care unit (ICU) immediately prior to surgery
* Pregnancy at the time of surgery
* Subsequent surgeries after index surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-13 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Amount of opioid medication used 72 hours post-extubation | From hospital admission for surgery to 72 hours after the patient is extubated postoperatively
  Opioid medication used at 72 hours post-extubation will be reported in morphine milligram equivalents

SECONDARY OUTCOMES:
Amount of opioid medication used 24 hours post-extubation | From hospital admission for surgery to 24 hours after the patient is extubated postoperatively
  Opioid medication used at 24 hours post-extubation will be reported in morphine milligram equivalents
Amount of opioid medication used 48 hours post-extubation | From hospital admission for surgery to 48 hours after the patient is extubated postoperatively
  Opioid medication used at 48 hours post-extubation will be reported in morphine milligram equivalents
Amount of opioid medication required throughout hospitalization | From the time the patient is extubated until the time the patient leaves the hospital, approximately 10 days. Safety to leave the hospital is determined by the cardiac surgery team and can be several days after surgery or longer.
  Opioid medication required from extubation until hospital discharge will be reported in morphine milligram equivalents
Amount of opioid medication required prior to extubation | From arrival in the ICU until extubation, approximately 6 hours. Safety of extubation is determined by the intensive care unit team and usually occurs within several hours of ICU arrival, although this can be variable.
  Opioid medication required between the end of surgery and extubation will be documented in morphine milligram equivalents.
Pain scores after extubation | 6 hours, 12 hours, 24 hours, 48 hours, and 72 hours after extubation
  Pain will be assessed by nursing staff using a numerical rating scale from 0-10, with 0 being no pain and 10 being the worst pain imaginable.
Time to extubation | From the time the patient arrives in the ICU intubated until the time they are successfully extubated, approximately 12 hours. Safety of extubation is determined by the ICU team and usually occurs within several hours, although this can be variable.
  This outcome will monitor the time in minutes from when a patient arrives in the ICU to the time the breathing tube is removed (extubation).

CONTACTS AND LOCATIONS:
Overall Officials: Krishnan Ramanujan, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No